CLINICAL TRIAL: NCT00455442
Title: A Two-Week, Double-Blind, Placebo-Controlled Study of the Efficacy and Safety of Mifepristone in the Prevention of Olanzapine-Induced Weight Gain in Healthy Male Volunteers
Brief Title: A Two-Week Study of the Efficacy and Safety of Mifepristone in the Prevention of Olanzapine-Induced Weight Gain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Collaborators: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: C-1073-200
Record Dates: First submitted 2007-03-30; First posted 2007-04-03 (Estimated); Last update posted 2008-09-19 (Estimated); Status verified 2008-09

CONDITIONS: Weight-Gain Prevention
MeSH Terms: interventions — Mifepristone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Mifepristone

SUMMARY:
This is a two-week study testing the efficacy and safety of mifepristone in the prevention of olanzapine-induced weight gain in healthy male volunteers by measuring changes in body weight and BMI.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers between 18 and 40 years of age
* BMI between ≥ 18 and ≤ 25
* Able to provide written informed consent
* Routine clinical laboratory tests either within normal limits or not clinically meaningful if outside of normal limits

Exclusion Criteria:

* History of Cushing's syndrome or Addison's disease
* Prior or current history of any psychiatric disorder, including eating disorders such as anorexia nervosa, bulimia nervosa, or binge-eating disorder
* Positive urine drug screen for any non-prescribed drug of abuse (including but not limited to amphetamines, cannabinoids, barbiturates, cocaine, opiates, benzodiazepines)
* Participation in a clinical investigation of any drug, biological or other investigational therapy within 30 days prior to dosing
* Have a history of an allergic reaction to either mifepristone or olanzapine
* Any clinically significant abnormality on screening laboratory tests
* QTc Bazzett's ≥ 450 msec
* Any major medical condition, which in the opinion of the Investigator would place the patient at undue risk.
* Receiving any prescription or over-the-counter medications that could potentially affect appetite or weight
* History of recent (within 6 months of screening) significant weight fluctuation

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2007-03; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
To determine the efficacy of mifepristone in the prevention of olanzapine-induced weight gain in healthy male volunteers.

SECONDARY OUTCOMES:
To determine the tolerability and safety of the administration of mifepristone and olanzapine in healthy male volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Thad Block, MD, Study Director — Corcept Therapeutics
Locations (1):
- St. John's Medical College, Bangalore, India

REFERENCES:
- [Background] Beebe KL, Block T, Debattista C, Blasey C, Belanoff JK. The efficacy of mifepristone in the reduction and prevention of olanzapine-induced weight gain in rats. Behav Brain Res. 2006 Aug 10;171(2):225-9. doi: 10.1016/j.bbr.2006.03.039. Epub 2006 Jun 19. PMID 16782211
- See also: Corcept Therapeutics official website — http://www.corcept.com